CLINICAL TRIAL: NCT05158062
Title: Phase II Study of Pembrolizumab and Bevacizumab in Combination With Platinum-based Chemotherapy Followed by Pembrolizumab, Bevacizumab and Olaparib in Patients With Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: Pembrolizumab and Bevacizumab With Chemotherapy Followed by Pembrolizumab, Bevacizumab and Olaparib in Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kosei Hasegawa, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Kosei Hasegawa, MD, PhD, Professor and Director, Department of Gynecologic Oncology, Saitama Medical University International Medical Center
Organization: Saitama Medical University International Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SaINT-ov02
Record Dates: First submitted 2021-11-26; First posted 2021-12-15 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Ovarian Epithelial
Keywords: ovarian cancer, pembrolizumab, olaparib
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — pembrolizumab; olaparib; Bevacizumab; Carboplatin; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- pembrolizumab and bevacizumab with PBC followed by pembrolizumab, bevacizumab and olaparib (Experimental): Participants will continue treatment period up to 6 cycles and enter maintenance period after treatment period. Study treatment will be continued until progressive disease (PD) based on RECIST 1.1, death, unacceptable toxicity, or participant withdrawal from the study.
  Interventions: Biological: pembrolizumab; Drug: olaparib; Biological: bevacizumab; Drug: carboplatin; Drug: paclitaxel; Drug: docetaxel

INTERVENTIONS:
Biological: pembrolizumab — pembrolizumab 200 mg every three weeks (Q3W)
  Other Names: KEYTRUDA
Drug: olaparib — olaparib 300 mg twice daily (BID) during maintenance period
  Other Names: LYNPARZA
Biological: bevacizumab — bevacizumab 15 mg/kg Q3W
  Other Names: AVASTIN
Drug: carboplatin — carboplatin AUC=5 or 6 Q3W during treatment period
Drug: paclitaxel — paclitaxel 175 mg/m2 Q3W during treatment period
Drug: docetaxel — docetaxel 60 ~ 70 mg/m2 Q3W during treatment period

SUMMARY:
This trial is a multicenter, single-arm, phase II study evaluating the efficacy of pembrolizumab and bevacizumab in combination with platinum-based chemotherapy (PBC) followed by pembrolizumab, bevacizumab and olaparib as a maintenance therapy in patients with platinum-sensitive recurrent ovarian cancer.This study is planned to enroll eligible 35 patients from multiple study sites in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is at least 20 years of age on the day of signing informed consent with histologically confirmed epithelial ovarian cancer (excluding borderline ovarian tumor) excluding mucinous carcinoma.
2. Participant has received only one regimen of PBC (3 cycles or more) as prior therapy with clinical CR (determined by negative clinical examination and a normal CA-125 level).
3. Participant has documentation of progressive disease at least 6 months from completion of PBC (platinum-sensitive).
4. Participant with measurable disease based on RECIST 1.1 at screening
5. Participant is able to provide a core or excisional biopsy of a tumor for testing of PD-L1 status, etc.
6. Participant with Eastern Cooperative Oncology Group (ECOG) PS of 0 to 1 at the screening
7. Participant has a life expectancy of at least 12 weeks as determined by the investigators.
8. Participant has adequate organ function.

Exclusion Criteria:

1. A Women of Childbearing Potential (WOCBP) who has a positive urine pregnancy test at screening. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Participant has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
3. Participant has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to the first dose of study drug.
4. Participant has received prior radiotherapy within 2 weeks of the first dose of study drug.
5. Participant has received major surgery within 4 weeks prior to the first dose of study drug.
6. Participant has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
7. Participant is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study drug.
8. Participant has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Participant has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
10. Participant has known active CNS metastases and/or carcinomatous meningitis.
11. Participant has severe hypersensitivity (≥Grade 3) to the study treatment and/or any of its excipients.
12. Participant has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
13. Participant has a history of (non-infectious) pneumonitis/interstitial lung disease that required treatment with steroids or has current pneumonitis/interstitial lung disease.
14. Participant has an active infection requiring systemic therapy.
15. Participant has a known history of Human Immunodeficiency Virus (HIV) infection.
16. Participant has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
17. Participant has received colony-stimulating factors (granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 2 weeks prior to the first dose of study drug.
18. Participant has clinically serious cardiovascular/cerebrovascular diseases (eg, cerebrovascular accident/stroke [less than 6 month prior to enrollment], myocardial infarction [less than 6 month prior to enrollment], uncontrolled and potentially reversible cardiac conditions [unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 msec, electrolyte disturbances, hypertension defined as systolic >150 mmHg or diastolic >90 mmHg etc.] or participant has congenital long QT syndrome).
19. Participant has known abdominal fistula, gastrointestinal fistula or gastrointestinal perforation and/or higher risks of bleeding.
20. Participant has either myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or has features suggestive of MDS/AML.
21. Participant is currently receiving either strong (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate (eg, ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued prior to the first dose of study drug.
22. Participant is currently receiving either strong (eg, phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine, and St John's Wort) or moderate (eg, bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued prior to the first dose of study drug.
23. Participant is either unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (eg, gastrectomy, partial bowel obstruction, malabsorption).
24. Participant has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
25. Participant is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 210 days after the last dose of study treatment.
26. Participant has had an allogenic tissue/solid organ transplant.
27. Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the investigators.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Two-year progression-free survival rate | 2 years
  Two-year progression-free survival rate after administration of pembrolizumab and bevacizumab in combination with PBC followed by pembrolizumab, bevacizumab and olaparib as a maintenance therapy in patients with platinum-sensitive recurrent ovarian cancer based on RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 3 years
  PFS after administration of the study treatment based on RECIST 1.1
PFS in maintenance period by chemotherapy responder | 3 years
  PFS in maintenance period in patients who assessed CR or PR at last tumor assessment before entering maintenance period based on RECIST 1.1
Objective Response Rate (ORR) | 3 years
  ORR after administration of the study treatment based on RECIST 1.1
Disease Control Rate (DCR) | 3 years
  DCR after administration of the study treatment based on RECIST 1.1
Duration of Response (DOR) | 3 years
  DOR after administration of the study treatment based on RECIST 1.1
One-year progression-free survival rate | 1 year
  One-year progression-free survival rate after administration of the study treatment based on RECIST 1.1.
Overall Survival (OS) | 3 years
  OS after administration of the study treatment using Kaplan-Meier method
Incidence of adverse events | 3 years
  The number and proportion of participants with adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
Biomarkers | 3 years
  Exploratory assessment of relationship between biomarkers and efficacy endpoints if possible

CONTACTS AND LOCATIONS:
Overall Officials: Kosei Hasegawa, MD, PhD, Principal Investigator — Saitama Medical University International Medical Center
Locations (1):
- Saitama Medical Uiversity International Medical Center, Hidaka, Saitama, Japan

IPD SHARING:
Plan to Share IPD: No